CLINICAL TRIAL: NCT03589469
Title: A Phase 2 Open-Label Single-Arm Study to Evaluate the Efficacy and Safety of Loncastuximab Tesirine in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) (LOTIS-2)
Brief Title: Study to Evaluate the Efficacy and Safety of Loncastuximab Tesirine in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: LOTIS-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-201; 2017-004288-11 (EudraCT Number)
Record Dates: First submitted 2018-05-04; First posted 2018-07-18 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Diffuse Large B-Cell Lymphoma Refractory; Diffuse Large B-cell Lymphoma Recurrent
Keywords: Loncastuximab tesirine
MeSH Terms: interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Loncastuximab tesirine (Experimental): Participants will receive loncastuximab tesirine as an IV infusion over 30 minutes on Day 1 of each cycle (every 3 weeks) at a dose of 150 μg/kg Q3W for 2 cycles, then 75 μg/kg Q3W for subsequent cycles for up to one year or until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: Loncastuximab tesirine

INTERVENTIONS:
Drug: Loncastuximab tesirine — intravenous infusion
  Other Names: Zynlonta; ADCT-402

SUMMARY:
The purpose of this Phase 2 study is to evaluate the clinical efficacy and safety of Loncastuximab Tesirine (ADCT-402) in patients with relapsed or refractory Diffuse Large B-Cell Lymphoma.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, open-label, single-arm study of the efficacy and safety of loncastuximab tesirine used as monotherapy in patients with relapsed or refractory DLBCL. The study will enroll approximately 140 patients

Loncastuximab Tesirine is an antibody drug conjugate (ADC) composed of a humanized antibody directed against human cluster of differentiation 19 (CD19), stochastically conjugated through a cathepsin-cleavable linker to SG3199, a pyrrolobenzodiazepine (PBD) dimer cytotoxin. Loncastuximab tesirine has been designed to target and kill CD19-expressing malignant B-cells.

A 2-stage design will be used in this clinical study, with an interim analysis for futility on the first 52 patients. If ≥10 patients respond (CR+PR), the study will proceed to complete full enrollment. Enrollment will continue during the interim analysis; however, further enrollment will be halted if futility is confirmed.

For each patient, the study will include a Screening Period (of up to 28 days), a Treatment Period (cycles of 3 weeks), and a Follow-up Period (approximately every 12 week visits for up to 3 years after treatment discontinuation).

Patients may continue treatment until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years or older.
* Pathologic diagnosis of DLBCL, as defined by the 2016 WHO classification, to include: DLBCL not otherwise specified; primary mediastinal large B-cell lymphoma; and high-grade B-cell lymphoma, with MYC and BCL2 and/or BCL6 rearrangements
* Relapsed or refractory disease following two or more multi-agent systemic treatment regimens
* Patients who have received previous CD19-directed therapy must have a biopsy that shows CD19 protein expression after completion of the CD19-directed therapy.
* Measurable disease as defined by the 2014 Lugano Classification
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block or minimum 10 freshly cut unstained slides if block is not available
* ECOG performance status 0-2
* Adequate organ function
* Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to start of study drug (C1D1) for women of childbearing potential
* Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the last dose of loncastuximab tesirine. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the patient receives his last dose of loncastuximab tesirine.

Exclusion Criteria:

* Previous treatment with loncastuximab tesirine
* Known history of hypersensitivity to or positive serum human ADA to a CD19 antibody
* Pathologic diagnosis of Burkitt lymphoma
* Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary
* Autologous stem cell transplant (ASCT) within 30 days prior to start of study drug (C1D1)
* Allogeneic stem cell transplant (AlloSCT) within 60 days prior to start of study drug (C1D1)
* Active graft-versus-host disease
* Post-transplant lymphoproliferative disorders
* Active autoimmune disease, including motor neuropathy considered of autoimmune origin and other central nervous system (CNS) autoimmune disease
* Known seropositive and requiring anti-viral therapy for human immunodeficiency (HIV) virus, hepatitis B virus (HBV), or hepatitis C virus (HCV).
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis
* Lymphoma with active CNS involvement at the time of screening, including leptomeningeal disease
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* Breastfeeding or pregnant
* Significant medical comorbidities
* Major surgery, radiotherapy, chemotherapy or other anti-neoplastic therapy within 14 days prior to start of study drug (C1D1), except shorter if approved by the Sponsor
* Use of any other experimental medication within 14 days prior to start of study drug (C1D1)
* Planned live vaccine administration after starting study drug (C1D1)
* Failure to recover to Grade ≤1 (Common Terminology Criteria for Adverse Events version 4.0 [CTCAE v4.0]) from acute non-hematologic toxicity (Grade ≤2 neuropathy or alopecia) due to previous therapy prior to screening
* Congenital long QT syndrome or a corrected QTcF interval of >480 ms at screening (unless secondary to pacemaker or bundle branch block)
* Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the patient inappropriate for study participation or put the patient at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (24):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Compassionate Care Research Group, Inc., at Compassionate Care Medical Group, Inc., Fountain Valley, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University of Miami Hospital and Clinics, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC-Drug Shipment, Lab and Study Supplies Only, Marietta, Georgia
  - Medical Oncology & Hematology Associates, Des Moines, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center/ Nebraska Medicine, Omaha, Nebraska
  - North Shore Hematology Oncology Associates DBA NY Cancer and Blood Specialists, East Setauket, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - GHD Cancer Institute, Greenville, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Vista Oncology Inc. PS, Olympia, Washington
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Italy (5):
  - A.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Istituto di Ematologia Seragnoli, Bologna, BO
  - U.O. Oncologia ed Ematologia, Rozzano, Milano
  - Dipartimento di Oncomatlolgia - Unita Linfomi, Milan
  - Divisione di Oncoematologia, Milan
- Anastasios Stathis, Bellinzona, Canton Ticino, Switzerland
- United Kingdom (7):
  - University Hospitals of Leicester NHS Trust., Leicester, England
  - University College London Hospital, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Oxford Cancer Centre, Churchill Hospital, Oxford, England
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland
  - Abertawe Bro Morgannwg University Health Board - Singleton Hospital, Swansea, Wales
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuker RA, Alderuccio JP, Han S, Polar MK, Crane TE, Moskowitz CH, Yang F. Deep Learning-Based Body Composition Analysis for Outcome Prediction in Relapsed/Refractory Diffuse Large B-Cell Lymphoma: Insights From the LOTIS-2 Trial. JCO Clin Cancer Inform. 2025 Jul;9:e2500051. doi: 10.1200/CCI-25-00051. Epub 2025 Jul 16. PMID 40669032
- [Derived] Alderuccio JP, Reis IM, Hamadani M, Nachiappan M, Leslom S, Kahl BS, Ai WZ, Radford J, Solh M, Ardeshna KM, Hess BT, Lunning MA, Zinzani PL, Stathis A, Carlo-Stella C, Lossos IS, Caimi PF, Han S, Yang F, Kuker RA, Moskowitz CH. PET/CT Biomarkers Enable Risk Stratification of Patients with Relapsed/Refractory Diffuse Large B-cell Lymphoma Enrolled in the LOTIS-2 Clinical Trial. Clin Cancer Res. 2024 Jan 5;30(1):139-149. doi: 10.1158/1078-0432.CCR-23-1561. PMID 37855688
- [Derived] Caimi PF, Ai WZ, Alderuccio JP, Ardeshna KM, Hamadani M, Hess B, Kahl BS, Radford J, Solh M, Stathis A, Zinzani PL, Wang Y, Qin Y, Wang L, Xu ZC, Carlo-Stella C. Loncastuximab tesirine in relapsed/refractory diffuse large B-cell lymphoma: long-term efficacy and safety from the phase II LOTIS-2 study. Haematologica. 2024 Apr 1;109(4):1184-1193. doi: 10.3324/haematol.2023.283459. PMID 37646659
- [Derived] Hamadani M, Chen L, Song Y, Xu MK, Liao L, Caimi PF, Carlo-Stella C. Matching-adjusted Indirect Comparison of the Efficacy of Loncastuximab Tesirine Versus Treatment in the Chemoimmunotherapy Era for Relapsed/Refractory Diffuse Large B-cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2022 Aug;22(8):e738-e744. doi: 10.1016/j.clml.2022.04.006. Epub 2022 Apr 8. PMID 35513980
- [Derived] Hess B, Townsend W, Ai W, Stathis A, Solh M, Alderuccio JP, Ungar D, Liao S, Liao L, Khouri L, Zhang X, Boni J. Efficacy and Safety Exposure-Response Analysis of Loncastuximab Tesirine in Patients with B cell non-Hodgkin Lymphoma. AAPS J. 2021 Dec 10;24(1):11. doi: 10.1208/s12248-021-00660-3. PMID 34893942
- [Derived] Spira A, Zhou X, Chen L, Gnanasakthy A, Wang L, Ungar D, Curiel R, Liao L, Radford J, Kahl B. Health-Related Quality of Life, Symptoms, and Tolerability of Loncastuximab Tesirine in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2022 Mar;22(3):158-168. doi: 10.1016/j.clml.2021.09.001. Epub 2021 Sep 22. PMID 34690090
- [Derived] Caimi PF, Ai W, Alderuccio JP, Ardeshna KM, Hamadani M, Hess B, Kahl BS, Radford J, Solh M, Stathis A, Zinzani PL, Havenith K, Feingold J, He S, Qin Y, Ungar D, Zhang X, Carlo-Stella C. Loncastuximab tesirine in relapsed or refractory diffuse large B-cell lymphoma (LOTIS-2): a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):790-800. doi: 10.1016/S1470-2045(21)00139-X. Epub 2021 May 11. PMID 33989558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 28 study sites in Italy, Switzerland, the United Kingdom, and the United States from 01 August 2018 to 09 August 2022.
Groups:
- Loncastuximab Tesirine: Participants received loncastuximab tesirine as an intravenous (IV) infusion over 30 minutes on Day 1 of each cycle (every 3 weeks) at a dose of 150 μg/kg once every 3 weeks (Q3W) for 2 cycles, then 75 μg/kg Q3W for subsequent cycles for up to one year or until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurred first.
Period: Overall Study
Arm/Group | Loncastuximab Tesirine
Started | 145
Participants Received Treatment | 145
Completed | 11
Not Completed | 134
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 20
Not completed — Death | 97
Not completed — Lost to Follow-up | 8
Not completed — Miscellaneous | 1

BASELINE CHARACTERISTICS:
Population: All-treated population - all participants who received at least 1 dose of treatment.
Groups:
- Loncastuximab Tesirine: Participants received loncastuximab tesirine as an IV infusion over 30 minutes on Day 1 of each cycle (every 3 weeks) at a dose of 150 μg/kg Q3W for 2 cycles, then 75 μg/kg Q3W for subsequent cycles for up to one year or until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurred first.
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 132
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 130
  Race: Black or African American | 5
  Race: Asian | 3
  Race: American Indian or Alaskan Native | 1
  Race: Native Hawaiian or Pacific Islander | 1
  Race: Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59
  United Kingdom | 31
  Italy | 53
  Switzerland | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR, as determined by central review according to the 2014 Lugano classification, defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR).
Time Frame: Up to 21.5 months
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
percentage of participants | 48.3 [39.9 to 56.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the time from the first documentation of tumor response to disease progression or death.
Time Frame: Up to 39 months
Population: Participants in the all-treated population who achieved a complete response (CR) or partial response (PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 70
months | 13.37 [6.87 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events.

3. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate defined as the percentage of treated participants with a best overall response (BOR) of CR.
Time Frame: Up to 39 months
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
percentage of participants | 24.8 [18.0 to 32.7]

4. Secondary Outcome: Relapse-free Survival (RFS)
Description: RFS was defined as the time from the documentation of CR to disease progression or death.
Time Frame: Up to 39 months
Population: Participants in the all-treated population who achieved CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 36
months | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events.

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time between start of treatment and the first documentation of recurrence, progression, or death.
Time Frame: Up to 40 months
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
months | 4.93 [2.89 to 8.31]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the start of treatment and death from any cause.
Time Frame: Up to 43 months
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
months | 9.53 [6.74 to 11.47]

7. Secondary Outcome: Number of Participants Who Experience Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that did not necessarily have to have a causal relationship with treatment. A TEAE was an adverse event with an onset that began or worsened on or after the first dose date and until 30 days after the last dose date, or start of a new anticancer therapy/procedure, whichever came earlier. TEAE assessments also included those per the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 Grade ≥3 AEs and serious TEAEs.
  AEs were graded using CTCAE version 4 and according to the following: Grade 1 = mild AE, Grade 2 = Moderate AE, Grade 3 = a severe AE, Grade 4 = life-threatening AE, and Grade 5 = death due to AE. For events not listed in the CTCAE criteria, the same grading was used.
Time Frame: Up to 599 days
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Participants
  Any TEAE | 143
  Grade ≥3 TEAE | 107
  Serious TEAE | 57

8. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Tests
Description: Clinical laboratory tests included hematology and chemistry. Clinically significant changes were determined by the Investigator.
Time Frame: Baseline up to 599 days
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Participants | 83

9. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital sign measurements included arterial blood pressure, heart rate, respiratory rate, and body temperature. Clinical significance was determined by the investigator.
Time Frame: Baseline up to 599 days
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Participants | 0

10. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline and End of Treatment
Description: ECOG (Eastern Cooperative Oncology Group) Performance Status is scored on a 6-point scale where higher scores indicate a worse outcome. ECOG scores include the following:
  * 0 = fully active, able to carry on all pre-disease performance without restriction
  * 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 = ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  * 3 = capable of only limited self-care; confined to bed or chair more than 50% of waking hours
  * 4 = completely disabled; cannot carry on any self-care; totally confined to bed or chair
  * 5 = dead
Time Frame: Baseline and end of treatment (up to 599 days)
Population: All-treated population - all participants who received at least 1 dose of treatment. Results are presented for participants with data available for analysis at end of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Participants
  Baseline: ECOG score 0 | 58
  Baseline: ECOG score 1 | 78
  Baseline: ECOG score 2 | 9
  Baseline: ECOG score 3 | 0
  Baseline: ECOG score 4 | 0
  Baseline: ECOG score 5 | 0
  End of treatment: number analyzed (Participants) | 111
  End of treatment: ECOG score 0 | 44
  End of treatment: ECOG score 1 | 50
  End of treatment: ECOG score 2 | 14
  End of treatment: ECOG score 3 | 2
  End of treatment: ECOG score 4 | 1
  End of treatment: ECOG score 5 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiograms (ECGs)
Description: Clinically significant changes from baseline for 12-lead ECGs were measured as abnormal QT interval corrected by Fridericia formula (QTcF) and QT interval corrected by Bazett formula (QTcB) values.
Time Frame: Baseline up to 599 days
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Participants
  QTcB maximum change from baseline: >30, <=60 msec | 30
  QTcB maximum change from baseline: >60 msec | 4
  QTcF maximum change from baseline: >30, <=60 msec | 23
  QTcF maximum change from baseline: >60 msec | 1

12. Secondary Outcome: Maximum Concentration (Cmax) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose and end of infusion
Population: Pharmacokinetic (PK) population: All participants in the per-protocol population (all participants in the all-treated population without major protocol deviations) with at least 1 pre-Cycle 1 Day 1 and 1 post-dose valid assessment. Only participants with data available for analysis are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 142
ng/mL
  Conjugated Antibody Cycle 1 | 2430 (38.8)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 117
  Conjugated Antibody Cycle 2 | 2734 (35.8)
  Conjugated Antibody Cycle 3: number analyzed (Participants) | 83
  Conjugated Antibody Cycle 3 | 1694 (47.6)
  Total Antibody Cycle 1 | 3267 (36.7)
  Total Antibody Cycle 2: number analyzed (Participants) | 117
  Total Antibody Cycle 2 | 3756 (31.3)
  Total Antibody Cycle 3: number analyzed (Participants) | 81
  Total Antibody Cycle 3 | 2581 (41.9)
  SG3199 Cycle 1: number analyzed (Participants) | 8
  SG3199 Cycle 1 | 0.0410 (56.6)
  SG3199 Cycle 2: number analyzed (Participants) | 5
  SG3199 Cycle 2 | 0.0490 (78.8)
  SG3199 Cycle 3: number analyzed (Participants) | 3
  SG3199 Cycle 3 | 0.0320 (20.3)

13. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose
Population: PK population: All participants in the per-protocol population (all participants in the all-treated population without major protocol deviations) with at least 1 pre-Cycle 1 Day 1 and 1 post-dose valid assessment. Only participants with data available for analysis are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 143
day*ng/mL
  Conjugated Antibody Cycle 1 | 15850 (105)
  Conjugated Antibody Cycle 2: number analyzed (Participants) | 116
  Conjugated Antibody Cycle 2 | 23913 (67.1)
  Conjugated Antibody Cycle 3: number analyzed (Participants) | 0
  Total Antibody Cycle 1 | 22160 (106)
  Total Antibody Cycle 2: number analyzed (Participants) | 116
  Total Antibody Cycle 2 | 33762 (67.2)
  Total Antibody Cycle 3: number analyzed (Participants) | 0
  SG3199 Cycle 1: number analyzed (Participants) | 8
  SG3199 Cycle 1 | 0.00400 (576)
  SG3199 Cycle 2: number analyzed (Participants) | 5
  SG3199 Cycle 2 | 0.00100 (204)
  SG3199 Cycle 3: number analyzed (Participants) | 0

14. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-∞) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 99
day*ng/mL
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 32
  Conjugated Antibody Cycle 1 | 19825 (52.9)
  Conjugated Antibody Cycle 2 | 26902 (33.4)
  Conjugated Antibody Cycle 3: number analyzed (Participants) | 0
  Total Antibody Cycle 1: number analyzed (Participants) | 27
  Total Antibody Cycle 1 | 25778 (61.3)
  Total Antibody Cycle 2: number analyzed (Participants) | 97
  Total Antibody Cycle 2 | 37761 (30.4)
  Total Antibody Cycle 3: number analyzed (Participants) | 0
  SG3199 Cycle 1: number analyzed (Participants) | 0
  SG3199 Cycle 2: number analyzed (Participants) | 0
  SG3199 Cycle 3: number analyzed (Participants) | 0

15. Secondary Outcome: Apparent Terminal Half-life (Thalf) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 90
days
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 32
  Conjugated Antibody Cycle 1 | 8.85 (53.5)
  Conjugated Antibody Cycle 2 | 15.2 (31.7)
  Conjugated Antibody Cycle 3: number analyzed (Participants) | 0
  Total Antibody Cycle 1: number analyzed (Participants) | 27
  Total Antibody Cycle 1 | 8.66 (54.6)
  Total Antibody Cycle 2: number analyzed (Participants) | 63
  Total Antibody Cycle 2 | 20.9 (56.5)
  Total Antibody Cycle 3: number analyzed (Participants) | 0
  SG3199 Cycle 1: number analyzed (Participants) | 0
  SG3199 Cycle 2: number analyzed (Participants) | 0
  SG3199 Cycle 3: number analyzed (Participants) | 0

16. Secondary Outcome: Apparent Clearance (CL) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose
Population: Pharmacokinetic (PK) population: All participants in the per-protocol population (all participants in the all-treated population without major protocol deviations) with at least 1 pre-Cyle 1 Day 1 and 1 post-dose valid assessment. Only participants with data available for analysis are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 99
L/day
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 32
  Conjugated Antibody Cycle 1 | 0.458 (47.6)
  Conjugated Antibody Cycle 2 | 0.331 (32.0)
  Total Antibody Cycle 1: number analyzed (Participants) | 27
  Total Antibody Cycle 1 | 0.418 (56.5)
  Total Antibody Cycle 2: number analyzed (Participants) | 97
  Total Antibody Cycle 2 | 0.285 (31.3)
  SG3199 Cycle 1: number analyzed (Participants) | 0
  SG3199 Cycle 2: number analyzed (Participants) | 0

17. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 90
liters
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 32
  Conjugated Antibody Cycle 1 | 4.24 (39.6)
  Conjugated Antibody Cycle 2 | 6.40 (36.5)
  Conjugated Antibody Cycle 3: number analyzed (Participants) | 0
  Total Antibody Cycle 1: number analyzed (Participants) | 27
  Total Antibody Cycle 1 | 4.10 (36.4)
  Total Antibody Cycle 2: number analyzed (Participants) | 63
  Total Antibody Cycle 2 | 7.54 (58.9)
  Total Antibody Cycle 3: number analyzed (Participants) | 0
  SG3199 Cycle 1: number analyzed (Participants) | 0
  SG3199 Cycle 2: number analyzed (Participants) | 0
  SG3199 Cycle 3: number analyzed (Participants) | 0

18. Secondary Outcome: Accumulation Index (AI) of Loncastuximab Tesirine Conjugated Antibody, Total Antibody and Warhead SG3199
Description: AI is the ratio of AUC0-last for each cycle divided by AUC0-last of the previous cycle.
Time Frame: Cycles 1 and 2: Day 1 pre-dose, and at 0, 4, 168 and 336 hours post-dose; Cycle 3: Day 1 pre-dose
Population: Pharmacokinetic (PK) population: All participants in the per-protocol population (all participants in the all-treated population without major protocol deviations) with at least 1 pre- Cyle 1 Day 1 and 1 post-dose valid assessment. Only participants with data available for analysis are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 90
ratio
  Conjugated Antibody Cycle 1: number analyzed (Participants) | 0
  Conjugated Antibody Cycle 2 | 1.65 (18.5)
  Conjugated Antibody Cycle 3: number analyzed (Participants) | 0
  Total Antibody Cycle 1: number analyzed (Participants) | 0
  Total Antibody Cycle 2: number analyzed (Participants) | 63
  Total Antibody Cycle 2 | 2.07 (38.1)
  Total Antibody Cycle 3: number analyzed (Participants) | 0
  SG3199 Cycle 1: number analyzed (Participants) | 0
  SG3199 Cycle 2: number analyzed (Participants) | 0
  SG3199 Cycle 3: number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants With an Anti-drug Antibody (ADA) Response to Loncastuximab Tesirine
Time Frame: Up to 599 days
Population: All-treated population - all participants who received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 145
Participants
  Confirmed Positive ADA Pre-dose | 1
  Confirmed Positive ADA Post-dose Only | 0
  Confirmed Positive ADA Anytime | 1

20. Secondary Outcome: Change From Baseline Score in the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: EQ-5D-5L is designed as an international, standardized, instrument for describing and evaluating quality of life (QoL). In the EQ-5D-5L VAS participants are asked to indicate their health state today on a VAS with the endpoints labeled 'the best health you can imagine' (score 100) and 'the worst health you can imagine' (score 0).
  A higher score on the VAS indicates better health related QoL. A positive change from baseline indicates an improvement in health related QoL.
Time Frame: Baseline, Day 1 of Cycles 2 to 26 (cycle duration of 3 weeks), and end of treatment (up to 599 days)
Population: Patient reported outcome (PRO) population. Only participants with data available for analysis are included. Overall number of participants analyzed prepresents all participants who contributed data to this assessment, though not all participants contributed data to each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 130
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 108
  Cycle 2 Day 1 | -0.1 (15.97)
  Cycle 3 Day 1: number analyzed (Participants) | 76
  Cycle 3 Day 1 | 1.3 (16.85)
  Cycle 4 Day 1: number analyzed (Participants) | 58
  Cycle 4 Day 1 | 2.8 (15.00)
  Cycle 5 Day 1: number analyzed (Participants) | 44
  Cycle 5 Day 1 | 2.8 (13.50)
  Cycle 6 Day 1: number analyzed (Participants) | 33
  Cycle 6 Day 1 | 3.0 (17.45)
  Cycle 7 Day 1: number analyzed (Participants) | 28
  Cycle 7 Day 1 | 4.0 (12.91)
  Cycle 8 Day 1: number analyzed (Participants) | 22
  Cycle 8 Day 1 | 7.3 (12.87)
  Cycle 9 Day 1: number analyzed (Participants) | 20
  Cycle 9 Day 1 | 7.7 (15.69)
  Cycle 10 Day 1: number analyzed (Participants) | 13
  Cycle 10 Day 1 | 12.2 (15.64)
  Cycle 11 Day 1: number analyzed (Participants) | 12
  Cycle 11 Day 1 | 11.8 (17.62)
  Cycle 12 Day 1: number analyzed (Participants) | 10
  Cycle 12 Day 1 | 16.3 (16.06)
  Cycle 13 Day 1: number analyzed (Participants) | 8
  Cycle 13 Day 1 | 6.0 (16.54)
  Cycle 14 Day 1: number analyzed (Participants) | 6
  Cycle 14 Day 1 | 12.2 (15.43)
  Cycle 15 Day 1: number analyzed (Participants) | 5
  Cycle 15 Day 1 | 6.6 (12.36)
  Cycle 16 Day 1: number analyzed (Participants) | 4
  Cycle 16 Day 1 | 5.5 (13.70)
  Cycle 17 Day 1: number analyzed (Participants) | 4
  Cycle 17 Day 1 | 8.3 (13.62)
  Cycle 18 Day 1: number analyzed (Participants) | 3
  Cycle 18 Day 1 | 11.0 (11.53)
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | 11.5 (16.26)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | 23.0 (NA) — Standard deviation could not be calculated as n = 1.
  Cycle 21 Day 1: number analyzed (Participants) | 2
  Cycle 21 Day 1 | 16.5 (9.19)
  Cycle 22 Day 1: number analyzed (Participants) | 2
  Cycle 22 Day 1 | 16.5 (9.19)
  Cycle 23 Day 1: number analyzed (Participants) | 1
  Cycle 23 Day 1 | 23.0 (NA) — Standard deviation could not be calculated as n = 1.
  Cycle 24 Day 1: number analyzed (Participants) | 1
  Cycle 24 Day 1 | 23.0 (NA) — Standard deviation could not be calculated as n = 1.
  Cycle 25 Day 1: number analyzed (Participants) | 1
  Cycle 25 Day 1 | 23.0 (NA) — Standard deviation could not be calculated as n = 1.
  Cycle 26 Day 1: number analyzed (Participants) | 1
  Cycle 26 Day 1 | 23.0 (NA) — Standard deviation could not be calculated as n = 1.
  End of treatment: number analyzed (Participants) | 98
  End of treatment | -8.3 (19.85)

21. Secondary Outcome: Change From Baseline Score in the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) - Lymphoma Subscale (LymS)
Description: Composed of the Functional Assessment of Cancer Therapy - General (FACT-G) plus the 15-item LymS. The FACT-G questionnaire contains 27 items covering 4 core health related quality of life (QoL) subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The LymS addresses issues including pain, itching, night sweats, trouble sleeping, fatigue and trouble concentrating. Score range for the LymS was 0 - 60, where a higher score indicates less symptoms. The LymS score is reported. A positive change from baseline indicates an improvement in health related QoL.
Time Frame: Baseline, Day 1 of Cycles 2 to 25 (cycle duration of 3 weeks), and end of treatment (up to 599 days)
Population: PRO population. Only participants with data available for analysis are included. Overall number of participants analyzed represents all participants who contributed data to this assessment, though not all participants contributed data to each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Loncastuximab Tesirine
Number analyzed (Participants) | 130
score on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 110
  Cycle 2 Day 1 | 0.95 (7.114)
  Cycle 3 Day 1: number analyzed (Participants) | 78
  Cycle 3 Day 1 | 1.34 (8.764)
  Cycle 4 Day 1: number analyzed (Participants) | 60
  Cycle 4 Day 1 | 2.09 (8.832)
  Cycle 5 Day 1: number analyzed (Participants) | 47
  Cycle 5 Day 1 | 0.16 (8.506)
  Cycle 6 Day 1: number analyzed (Participants) | 33
  Cycle 6 Day 1 | 1.16 (9.918)
  Cycle 7 Day 1: number analyzed (Participants) | 29
  Cycle 7 Day 1 | 1.00 (11.474)
  Cycle 8 Day 1: number analyzed (Participants) | 22
  Cycle 8 Day 1 | 3.43 (10.141)
  Cycle 9 Day 1: number analyzed (Participants) | 20
  Cycle 9 Day 1 | 2.17 (9.498)
  Cycle 10 Day 1: number analyzed (Participants) | 13
  Cycle 10 Day 1 | 3.18 (11.769)
  Cycle 11 Day 1: number analyzed (Participants) | 12
  Cycle 11 Day 1 | 4.35 (13.053)
  Cycle 12 Day 1: number analyzed (Participants) | 10
  Cycle 12 Day 1 | 4.90 (11.140)
  Cycle 13 Day 1: number analyzed (Participants) | 9
  Cycle 13 Day 1 | 2.01 (16.871)
  Cycle 14 Day 1: number analyzed (Participants) | 6
  Cycle 14 Day 1 | 0.63 (17.442)
  Cycle 15 Day 1: number analyzed (Participants) | 5
  Cycle 15 Day 1 | -3.27 (7.691)
  Cycle 16 Day 1: number analyzed (Participants) | 4
  Cycle 16 Day 1 | -8.04 (10.561)
  Cycle 17 Day 1: number analyzed (Participants) | 4
  Cycle 17 Day 1 | -6.88 (9.360)
  Cycle 18 Day 1: number analyzed (Participants) | 3
  Cycle 18 Day 1 | -5.00 (7.937)
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | -1.00 (4.243)
  Cycle 20 Day 1: number analyzed (Participants) | 2
  Cycle 20 Day 1 | -2.25 (4.596)
  Cycle 21 Day 1: number analyzed (Participants) | 2
  Cycle 21 Day 1 | -0.50 (2.121)
  Cycle 22 Day 1: number analyzed (Participants) | 2
  Cycle 22 Day 1 | -1.00 (2.828)
  Cycle 23 Day 1: number analyzed (Participants) | 1
  Cycle 23 Day 1 | 1.00 (NA) — Standard deviation could not be calculated as n = 1.
  Cycle 24 Day 1: number analyzed (Participants) | 0
  Cycle 25 Day 1: number analyzed (Participants) | 1
  Cycle 25 Day 1 | 1.00 (NA) — Standard deviation could not be calculated as n = 1.
  End of treatment: number analyzed (Participants) | 98
  End of treatment | -1.19 (9.042)

ADVERSE EVENTS:
Time Frame: Up to 43 months
Description: All non-serious AEs at a frequency threshold of >=5% and all SAEs, regardless of relationship to study drug, were reported from the time the participant signs the ICF until 30 days after the last dose of study drug or start of new anti-cancer therapy, whichever is earlier; thereafter, only related SAEs were collected, with two exceptions of participants with subsequent SCT or CAR-T therapy.
Arm/Group | Loncastuximab Tesirine
All-Cause Mortality (participants affected / at risk) | 97/145
Serious Adverse Events (participants affected / at risk) | 57/145
Other Adverse Events (participants affected / at risk) | 139/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Loncastuximab Tesirine (N=145)
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Disease progression (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Metapneumovirus infection (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Facial nerve disorder (Nervous system disorders) | 1
Psychomotor skills impaired (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Postoperative hypotension (Injury, poisoning and procedural complications) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Loncastuximab Tesirine (N=145)
Neutropenia (Blood and lymphatic system disorders) | 58
Thrombocytopenia (Blood and lymphatic system disorders) | 48
Anaemia (Blood and lymphatic system disorders) | 38
Leukopenia (Blood and lymphatic system disorders) | 21
Lymphopenia (Blood and lymphatic system disorders) | 11
Tachycardia (Cardiac disorders) | 11
Nausea (Gastrointestinal disorders) | 34
Diarrhoea (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 16
Fatigue (General disorders) | 40
Oedema peripheral (General disorders) | 28
Pyrexia (General disorders) | 25
Asthenia (General disorders) | 14
Gamma-glutamyltransferase increased (Investigations) | 61
Blood alkaline phosphatase increased (Investigations) | 29
Alanine aminotransferase increased (Investigations) | 22
Aspartate aminotransferase increased (Investigations) | 23
Weight increased (Investigations) | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 23
Decreased appetite (Metabolism and nutrition disorders) | 22
Hypokalaemia (Metabolism and nutrition disorders) | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 20
Hypocalcaemia (Metabolism and nutrition disorders) | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 8
Headache (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 19
Pruritus (Skin and subcutaneous tissue disorders) | 19
Erythema (Skin and subcutaneous tissue disorders) | 15
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Hypotension (Vascular disorders) | 10
Hypertension (Vascular disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after first multi-site publication or if no multi-site publication is made within 18 months of study completion/termination. The only disclosure restriction on PI is sponsor can review results comms. prior to public release and can embargo comms. regarding trial results for a period >60 but ≤180 days from time submitted to sponsor review. Sponsor can't require changes to the comms, extend embargo or require changes to comms, except removing confidential info that are not results

DOCUMENTS (2):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03589469/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT03589469/SAP_002.pdf